CLINICAL TRIAL: NCT00116077
Title: Dopamine Receptor Imaging in Mood Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050169; 05-M-0169
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-11-12

CONDITIONS: Mood Disorders; Depressive Disorder, Major; Bipolar Disorder
Keywords: PET; [C-11] NNC-112; [F-18] Fallypride; Dopamine Receptors; Mood Disorders; DA Receptors; Major Depressive Disorder; Bipolar Disorder; MDD; Bipolar Depression; Healthy Volunteer; HV
MeSH Terms: conditions — Mood Disorders; Depressive Disorder, Major; Bipolar Disorder

SUMMARY:
This study seeks to increase the understanding of dopamine receptor function in the brain during major depressive disorder and bipolar depression, as well as genetic changes that may be behind changes in those receptors' actions. Dopamine is a natural messenger in the brain, involved in reward, motivation, and mood.

Volunteers aged 18 to 55 who have primary major depressive disorder and those who have bipolar depression (20 in each group), who are not HIV positive and do not have AIDS, and who are not pregnant or breastfeeding may be eligible for this study.

A telephone interview will be held, for patients to answer standardized questions about psychiatric or medical symptoms they may have experienced during their lifetime. Those eligible for the study will undergo interviews and laboratory tests. A psychiatric interview and clinical assessment will collect various data. Patients will undergo the following procedures and tests:

* A brief neurological examination
* A one-minute electrocardiogram to measure electrical activity of the heart.
* Laboratory tests measuring several substances in the blood and urine.
* Pregnancy test.

A magnetic resonance imaging (MRI) scan will be done to create an image of the volunteer's brain structure. The technique of MRI uses a strong magnetic field and radio waves to obtain images of body organs and tissues. During the MRI scan, volunteers will lie still on a table that will slide into the scanner for 30 minutes and in some cases up to but no more than 90 minutes. Volunteers will be asked to lie as still as possible during the procedure. Then a PET system will create two images of brain blood flow-one of brain dopamine 1 receptor and one of dopamine 2/3 receptor binding. Volunteers will be given a radiotracer, a tiny amount of a drug that can be detected by a special camera in the PET scanner. A tiny flexible tube will be placed in the vein of one arm during each PET scan but during the MRI scan. Volunteers will be asked to lie still on the PET scanner table. A mask with large holes for eyes, ears, and mouth will be placed over the head, to keep the head from moving. After radiotracer injections are given, the PET scanner will create brain images. There may be two PET scanning sessions, each requiring about 3 hours of scanning. During only one of these there will be breaks. At the end of the scanning session, volunteers will be asked to drink several glasses of water and urinate immediately, to reduce radiation exposure to the bladder wall.

Genetic screening will help to enhance researchers' understanding of the role of dopamine receptors in depression. A small blood sample, about 2 tablespoons, will be collected, to isolate DNA from blood cells. Some of the blood samples or DNA may be stored for future studies, but those samples will remain coded, so participants will not be identified. This study will not have a direct benefit for participants. However, the results may provide knowledge to help people in the future. This study does involve compensation.

DETAILED DESCRIPTION:
The dopaminergic projections from the substantia nigra and the ventral tegmental area into the ventral striatum and medial prefrontal cortex (mPFC) play major roles in the neural processing underlying motivated behavior. Hypofunction of this system is hypothesized to underlie the anhedonia, psychomotor slowing and amotivation that characterize major depressive disorder (MDD; (Fibiger, 1991; Swerdlow and Koob, 1987). A variety of indirect evidence supports this hypothesis (Wilner, 1995) as: 1) Cerebrospinal fluid (CSF) concentrations of the DA metabolite, homovanillic acid, are reduced in nondelusional, depressives. 2) Dextroamphetamine (AMPH) improves mood in depressed patients, and direct DA receptor agonists (e.g. pramapaxil) and DA reuptake inhibitors (e.g. nomiphensine) exert antidepressant effects. 3) Many somatic antidepressant therapies enhance D(2/3) receptor sensitivity in limbic structures and/or increase interstitial DA concentrations in the mPFC and accumbens in rats. 4) Conditions in which DA is depleted increase the risk for developing major depression, and DA receptor antagonist administration produces dysphoria, avolition and fatigue in healthy humans.

In more direct assessments of DA receptor pharmacology, Suhara et al. (1992) reported an abnormal decrease in D1 receptor binding using [(11)C]SCH 23390 in the frontal cortex of bipolar subjects. However, [(11)C]SCH 23390 has some affinity for 5-HT(2) receptors in the frontal cortex (De Keyser et al.,1988) so the specificity of this result remains unclear. In contrast, [(11)C]NNC 112 is selective for D1 receptors and shows sufficient receptor selectivity to access D(1) receptor binding in the frontal cortex in mood disorders.

Previous studies of D(2) receptors using [(11)C]raclopride, [11C]NMSP and [(123)I]IBZM have been limited by the lack of sensitivity of those radioligands to receptors outside the striatum. Striatal D(2) receptor binding has been reported to be abnormally increased in psychotic bipolar subjects relative to both controls and non-psychotic bipolar subjects using [(11)C]NMSP (Pearlson et al., 1995) and unaltered in subjects with Major Depressive Disorder (MDD) compared to controls in two studies using [(123)I]IBZM (Klimke et al., 1999; Parsey et al., 2001). An increased basal ganglia-to-cerebellum ratio of D(2) receptor binding using [(123)I]IBZM has been reported in depressed MDD subjects compared to controls (D'Hanenen and Bossuyt, 1994; Ebert et al., 1996). SPECT imaging studies show that [(123)I]IBZM binding to striatal D(2/3) receptors is abnormally elevated in MDD. Although these studies were confounded by medication effects and small subject samples, because [(123)I]IBZM binding is sensitive to competition from endogenous DA, this abnormality could reflect reduced intrasynaptic DA levels in the striatum of MDD subjects.

The current study will address the limitations of the previous studies by characterizing D1 and D2 receptor binding in depression in extrastriatal, as well as striatal regions. PET measures of [11C]NNC 112 and [(18)F]fallypride binding to assess D(1) and D(2/3) receptor binding potential (BP), respectively, in unmedicated depressed subjects (part A). The 11C-Raclopride Bolus plus constant infusion (B/I) PET scan will assess D(2) receptor binding in vivo in the striatum while the subjects perform a monetary reward task, specifically designed to induce changes in the striatal dopaminergic transmission (part B).

The application of high resolution 3D PET and MRI-based region-of-interest analysis will permit specific assessment of abnormalities of the D(2/3) receptor system in currently depressed individuals with MDD and BD and of correlations with clinical ratings in ventral and dorsal striatum as well as in extrastriatal areas such as the amygdala, anterior cingulate cortex, medial prefrontal cortex and orbital cortex. Possible relationships of polymorphisms in the genes coding for elements of the dopaminergic system as well as the dopamine receptors being studied in MDD or BD with the level of binding detected will be investigated collecting preliminary data.

SPECIFIC AIMS

1. Assess D(1) receptor binding in BD subjects and performance on working memory and attention based tasks.

   Hypothesis 1a. D(1) receptor binding will be decreased in the frontal cortex and unaltered in the striatum of BD subjects compared to healthy controls.

   Hypothesis 1b. Working memory and attention task performance impairments will correlate with changes in binding levels.
2. Evaluate striatal and extrastriatal D(2/3) receptor binding, severity of depression, psychomotor retardation and anhedonia in depressed subjects with BD or MDD compared to healthy controls.

Hypothesis 2a. Baseline [(18)F]fallypride binding in the ventral striatum, amygdala, medial thalamus, orbital cortex and subgenual PFC will be increased in depressives relative to controls.

Hypothesis 2b. The ventral striatal D(2/3) receptor binding will correlate positively with ratings of anhedonia and depressed mood, and negatively with psychomotor performance speed.

Hypothesis 2c. Baseline [(11)C] raclopride binding in the ventral striatum will be increased in depressed patients and this increase will correlate negatively with the subjective evaluation of rewarding stimuli and mood.

Hypothesis 2d. The monetary reward task will induce a reduction of [(11)C] raclopride striatal binding, which will be larger in controls than in depressed patients and correlate negatively with anhedonia scores.

Secondary Aims: A. To explore differences in D(1) and D(2/3) receptor binding between MDD and BD subjects.

B. To investigate whether polymorphisms for the D(1) or the D(2/3) receptor gene may be associated with differences in receptor BP.

C. To assess the relationship between [11C]NNC binding to D(1) receptors and performance on working memory and attention based tasks from the CANTAB (Cambridge Cognition, UK), including the Rapid Visual Information Processing test (RVIP) the Spatial Working Memory test (SWM) and the Pattern Recognition Memory test (PRM).

ELIGIBILITY:
* INCLUSION CRITERIA:

The presence of inclusion and exclusion criteria will be established using both unstructured psychiatric interview with a psychiatrist and the Structured Clinical Interview for DSM-IV (SCID; (Williams et al., 1992). Family history of mental illness will be obtained using the Family Interview of Genetic Studies (Maxwell, 1982).

MDD Depressed Sample: Forty-six subjects (ages 18-55) male and female will be selected, with primary MDD currently depressed as defined by DSM-IV criteria for recurrent MDD.

Bipolar Depressed Sample: Forty subjects (ages 18-55) male and female will be selected who meet DSM-IV criteria for bipolar I or II disorder and are currently depressed, with HDRS score in the moderately-to-severely depressed range (greater than 18). Subjects may be inpatients or outpatients. Because effective treatment will not be discontinued for the purposes of this protocol, subjects will be identified who have never been treated or who have discontinued medication due to lack of efficacy, noncompliance, physician order or other reasons prior to study entry.

Healthy, Control Sample: Forty-six subjects (ages 18-55) male and female who have not met criteria for any major psychiatric disorder will be selected. From this large sample a control subject will be matched to each depressed subject for age, gender, handedness and stage of menstrual cycle. The control subjects will have no known first degree relatives with mood disorders.

EXCLUSION CRITERIA:

Subjects must not have taken antidepressant or other medications likely to alter monoamine neurochemistry or cerebrovascular function for at least 3 weeks (8 weeks for fluoxetine and for any drug with known anticholinergic effects) prior to scanning. Because effective medications will not be discontinued for the purposes of this study, subjects will be identified who have never been treated or who have discontinued medication due to lack of efficacy, noncompliance, physician order or other reasons prior to study entry. Subjects will be excluded if they: a) have had serious suicidal ideation or behavior in the previous two months, or b) psychosis, or c) medical or neurological illnesses (i.e. seizure disorder, a coma in past) likely to affect physiology or anatomy, d) a history of drug or alcohol abuse within 1 year or a lifetime history of alcohol or drug dependence (DSM IV criteria), e) are HIV positive or have AIDS, f)current pregnancy (documented by history and pregnancy testing prior to scanning), g) current breast feeding, h) general MRI exclusion criteria which include the subject having a pacemaker or significant claustrophobia.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2005-06-21; Study Completion 2010-11-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abi-Dargham A, Mawlawi O, Lombardo I, Gil R, Martinez D, Huang Y, Hwang DR, Keilp J, Kochan L, Van Heertum R, Gorman JM, Laruelle M. Prefrontal dopamine D1 receptors and working memory in schizophrenia. J Neurosci. 2002 May 1;22(9):3708-19. doi: 10.1523/JNEUROSCI.22-09-03708.2002. PMID 11978847
- [Background] Alheid GF, Heimer L. New perspectives in basal forebrain organization of special relevance for neuropsychiatric disorders: the striatopallidal, amygdaloid, and corticopetal components of substantia innominata. Neuroscience. 1988 Oct;27(1):1-39. doi: 10.1016/0306-4522(88)90217-5. PMID 3059226
- [Background] Allard P, Norlen M. Unchanged density of caudate nucleus dopamine uptake sites in depressed suicide victims. J Neural Transm (Vienna). 1997;104(11-12):1353-60. doi: 10.1007/BF01294736. PMID 9503281